CLINICAL TRIAL: NCT05614180
Title: Chronic Total Occlusive Lesions CMR Study
Acronym: CTO-CMR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lin Zhao (Other)
Responsible Party: Sponsor-Investigator, Lin Zhao, Associate director of cardiology department, Beijing Anzhen Hospital
Organization: Beijing Anzhen Hospital (Other)
Other Study IDs: KS2022056
Record Dates: First submitted 2022-11-05; First posted 2022-11-14 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Chronic Total Occlusion; Image; Revascularization
Keywords: Chronic Total Occlusion; Cardiac magnetic resonance; Revascularization
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Percutaneous coronary intervention — Patients with a diagnose of coronary chronic total occlusions will be treated by percutaneous coronary intervention, as indicated by the heart-team.

SUMMARY:
This registry will include consecutive patients presenting with at least one chronic total occlusion on coronary angiogram who will be treated by percutaneous coronary intervention in our center. All patients will undergo a non-invasive assessment for myocardial ischemia/viability using cardiac magnetic resonance (CMR) prior to revascularization therapy. Follow up CMR will be repeated in all participants after three months and one year. Additionally, clinical outcomes and quality of life will be evaluated at baseline and at follow-up. Primary objective of this study is to investigate the the reduction in ischemia (as evaluated by follow-up CMR) and the severity of angina according to clinical evaluation (including Seattle Angina Questionnaires [SAQ], Canadian Class Score[CCS] and 6-mins walking test).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Presence of at least one untreated CTO at basal angiography (defined as a total occlusion in any major coronary vessel or relevant side branches [reference vessel diameter ≥2.5mm or as judged by two independent interventional cardiologists], with TIMI 0 in the distal segment and at least 3 months old
* Patient has a clinical indication to perform CTO PCI
* Willing to participate and able to understand, read and sign the informed consent document.

Exclusion Criteria:

* CMR contraindications
* Contraindications to adenosine or dobutamine
* Severe chronic kidney disease (estimated Glomerular Filtration Rate [eGFR] <60 mL/min/1.73m2 or serum creatinine level >2.5 mg/dL)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients presenting with a diagnose of coronary chronic total occlusions undergoing percutaneous coronary intervention.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in ischemia | 3 months; 12 months
  Parameters of cardiac magnetic resonance

SECONDARY OUTCOMES:
Rate of target lesion failure (TLF). | 12 months
  TLF is defined as a composite of: cardiac death, target vessel myocardial infarction (SCAI definition), and clinically driven TLR.
Changes in angina paramteres | 3 months; 12 months
  Parameters of angina questionnaires.
Change of left ventricular structure and function | 3 months; 12 months
  Parameters of left ventricular function and structure on cardiac magnetic resonance

CONTACTS AND LOCATIONS:
Overall Officials: Lin Zhao, MD, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing anzhen hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No